CLINICAL TRIAL: NCT03129724
Title: Retrospective Study in Patients With Metastatic Renal Cancer Treated With TKI Sequence (Tyrosine Kinase Inhibitors of VEGFR) - mTOR- Axitinib Inhibitors or Anti-VEGF Antibody -Inhibiteurs mTOR - Axitinib
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6154
Record Dates: First submitted 2016-07-05; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2016-07

CONDITIONS: Kidney Neoplasms
Keywords: Kidney Neoplasms; Kidney; Neoplasms; TKI; Axitinib; VEGF; mTORi
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Describe in patients with metastatic kidney cancer treatment modalities with the type sequences: TKI - mTORi - Axitinib or VEGF mAb - mTORi - Axitinib.

ELIGIBILITY:
Inclusion criteria:

* Patient with metastatic kidney cancer (all histological types)
* Male or female aged (e) of 18 or more
* Patient has been treated or under treatment with axitinib (Inlyta®) in the third line after the first line of targeted TKI therapy and after mTORi in 2nd line, or
* Patient receiving the treatment sequence VEGFmAb - mTORi - axitinib For living patients: patient informed and having given oral consent

Exclusion criteria:

* Patient who received more than one line of antiangiogenic therapy in the metastatic phase before initiation of treatment with axitinib (except patients in the study Pisces) Patient received a second line treatment with TKI Patient refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with metastatic kidney cancer (all histological types) Patient has been treated or under treatment with axitinib (Inlyta®) in the third line after the first line of targeted TKI therapy and after mTORi in 2nd line, or Patient receiving the treatment sequence VEGFmAb - mTORi - axitinib
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of Kidney cancer | after surgery, up to 1 year]

IPD SHARING:
Plan to Share IPD: No